CLINICAL TRIAL: NCT00964652
Title: Treadmill Training With Additional Body Load: Effects on Gait of Subjects With Parkinson´s Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Nadiesca Taisa Filippin, Universidade Federal de Sao Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 234/2007
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Parkinson´s Disease
Keywords: treadmill; body load; Parkinson's disease; gait
MeSH Terms: conditions — Parkinson Disease

ARMS (1):
- PD Group (Experimental): Nine subjects with idiopathic PD, previously diagnosed by one specialist physician participated in this study.
  Interventions: Other: Treadmill walking training with additional body load

INTERVENTIONS:
Other: Treadmill walking training with additional body load — The training program was divided into three phases (A1-B-A2):
  treadmill training with additional body load (A1), control condition (conventional physical therapy) (B). and treadmill training with additional body load again (A2). Each phase lasted six weeks, totaling 18 weeks. Both evaluations and training were performed during on-phase of the medication cycle.

SUMMARY:
Background: Studies about the effects of walking training with additional body load in Parkinson's disease (PD) are lacking. There is evidence that the increase of body load during treadmill walking improves reflex activity and leg extensor muscle activity, which are impaired in subjects with PD.

Purpose: The purpose of this study was to assess the effects of treadmill walking training with additional body load on the ground reaction forces, spatiotemporal, and kinematic variables of the gait of subjects with moderate PD.

Design: This study was an A1-B-A2 single-case. Setting: The evaluation and the training were conducted in a movement analysis laboratory, and at the rehabilitation unit of the University, respectively.

Participants: Nine patients with PD (Hoehn and Yahr 2 through 3) and gait disturbances.

Interventions: Phases A1 and A2 included 6 weeks of gait training on a treadmill with 10% increase of normal body mass. Phase B included 6 weeks of conventional physical therapy.

Measurements: Measures included the ground reaction forces, spatiotemporal, and kinematic variables during overground walking, at baseline and after each phase.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD (previously diagnosed by one specialist physician,)
* Hoehn and Yahr (H-Y) stages 2 through 3,
* Absence of dementia (Mini-Mental Status Examination - MMSE, defined according to educational level) and,
* Capacity to ambulate independently for at least 10 meters.

Exclusion Criteria:

* Change medication (dopaminergic) during the study period,
* Use treadmill for at least six months prior to the study, and
* Other neurologic problems or musculoskeletal, cardiovascular and respiratory disease or uncorrected visual deficit that could represent risk and interfere in the performance of the training.

Ages: 51 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Significant increase in propulsive forces, stride length, speed, maximum hip extension during stance were observed after the training program. | 4 times, once before treatment, and 3 after each treatment phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil